CLINICAL TRIAL: NCT04039308
Title: Assessment of Surgical Correction of Deformity in Diabetic Charcot Arthropathy of the Foot and Ankle
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kerolos Maged (Other)
Responsible Party: Sponsor-Investigator, Kerolos Maged, Resident of Orthopedics and traumatology, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Deformity in Charcot foot
Record Dates: First submitted 2019-07-19; First posted 2019-07-31 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Deformity, Foot
MeSH Terms: conditions — Foot Deformities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The surgical techniques described in the literature for surgical management of diabetic charcot arthropathy of the foot and ankle include simple exostectomy, open reduction and internal fixation of neuropathic fractures, external fixation, arthrodesis, Achilles tendon lengthening. Patients are followed up at 1 year postoperative by an x-ray of the foot and ankle anteroposterior , lateral and oblique views to assess rate of union ,the correction of deformity by measuring the foot angles . The functional outcome is assessed by the AOFAS scoring system and the diabetic foot ulcer scaoeuulcer scale(18).

DETAILED DESCRIPTION:
Diabetes mellitus affected approximately 422 million people worldwide in 2016 . Diabetic complications including diabetic peripheral neuropathy and peripheral arterial disease remain prevalent in the USA and worldwide and challenging to treat. Due to loss of protective sensation and impaired vascular supply, these can lead to serious foot complications including deformity, diabetic foot ulceration, Charcot neuroarthropathy and infection .

Charcot neuroarthropathy is a devastating orthopedic condition that afflicts patients with diabetes. It is an inflammatory condition that affects the foot and ankle with varying degrees of bone destruction and deformity. The true incidence or prevalence of this condition is not known.

However, estimates demonstrate incidence to be between 0.1 and 0.9%

. Two principal pathways for the disease have been proposed. The neurotraumatic theory suggests that the loss of neuroprotection causes repetitive microtrauma. The opposing hypothesis, the neurovascular, is that sympathetic neuropathy results in hyperaemia. This leads to increased osteoclastic activity resulting in bone resorption and fragmentation.

The active form of charcot foot arthropahy is often misdiagnosed as tenosynovitis, cellulitis, or gout. The majority of these patients endure a short period of disability that is treated by some form of immobilization for a variable period of time with minimal resultant long-term disability. The diagnosis is not often clear until resolution of the swelling when a resultant residual deformity is appreciated.

Eichenholtz classification is used to define Charcot foot clinical stages. Brodsky the classification, in the other hand, allows us to locate the lesion anatomically.

The incidence of diabetic neuroarthropathy varies among the anatomical regions of the foot and ankle according to Brodsky classification. Approximately 70% of cases affect the tarsometatarsal joint (type 1). Type-1 disease is the least likely to require surgical stabilization, although the most common type to cause plantar ulceration. Type-2 disease involves the midtarsal and subtalar joints and accounts for approximately 20% of cases. Type-3 disease affects approximately 10% of patients, and occurs mainly in the ankle. Type 2 and type 3 are the most likely to progress to instability and often require long-term bracing or surgical reconstruction.

The surgical techniques described in the literature include simple exostectomy, open reduction and internal fixation of neuropathic fractures, external fixation, arthrodesis, Achilles tendon lengthening and, eventually, amputation.The goal of Charcot neuroarthropathy treatment, both orthopedic and surgical is to obtain an ulcer free, stable plantigrade foot, without osteomyelitis and able to ambulate. Achieving these goals notably reduces the rate of amputations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inactive form of Charcot arthropathy of the foot and ankle due to diabetes mellitus.

Patients received surgical management.

Exclusion Criteria:

* Active form of Charcot arthropathy of the foot and ankle. Non deforming Charcot arthropathy of the foot and ankle. Patients with heavy infection or vascular affection that necessitate amputation.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with deforming Charcot neuroarthropathy of the foot and ankle
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of postoperative deformity correction in at least one- year postoperative follow up1x rays. | 3 years
  Assessment of accuracy of correction in patients with Charcot neuroarthropathy of the foot and ankle using follow up x rays and measuring the foot and ankle angles. The normal angles are documented, so we will compare these angles with the normal ones.

REFERENCES:
- [Background] 1-World Health Organzation, Global report on diabetes .Geneva 2016
- [Background] Pop-Busui R, Boulton AJ, Feldman EL, Bril V, Freeman R, Malik RA, Sosenko JM, Ziegler D. Diabetic Neuropathy: A Position Statement by the American Diabetes Association. Diabetes Care. 2017 Jan;40(1):136-154. doi: 10.2337/dc16-2042. No abstract available. PMID 27999003
- [Background] Rogers LC, Frykberg RG, Armstrong DG, Boulton AJ, Edmonds M, Van GH, Hartemann A, Game F, Jeffcoate W, Jirkovska A, Jude E, Morbach S, Morrison WB, Pinzur M, Pitocco D, Sanders L, Wukich DK, Uccioli L. The Charcot foot in diabetes. Diabetes Care. 2011 Sep;34(9):2123-9. doi: 10.2337/dc11-0844. PMID 21868781
- [Background] Lavery LA, Armstrong DG, Wunderlich RP, Tredwell J, Boulton AJ. Diabetic foot syndrome: evaluating the prevalence and incidence of foot pathology in Mexican Americans and non-Hispanic whites from a diabetes disease management cohort. Diabetes Care. 2003 May;26(5):1435-8. doi: 10.2337/diacare.26.5.1435. PMID 12716801
- [Background] Prompers L, Schaper N, Apelqvist J, Edmonds M, Jude E, Mauricio D, Uccioli L, Urbancic V, Bakker K, Holstein P, Jirkovska A, Piaggesi A, Ragnarson-Tennvall G, Reike H, Spraul M, Van Acker K, Van Baal J, Van Merode F, Ferreira I, Huijberts M. Prediction of outcome in individuals with diabetic foot ulcers: focus on the differences between individuals with and without peripheral arterial disease. The EURODIALE Study. Diabetologia. 2008 May;51(5):747-55. doi: 10.1007/s00125-008-0940-0. Epub 2008 Feb 23. PMID 18297261
- [Background] El-Mowafi H, Abulsaad M, Kandil Y, El-Hawary A, Ali S. Hybrid Fixation for Ankle Fusion in Diabetic Charcot Arthropathy. Foot Ankle Int. 2018 Jan;39(1):93-98. doi: 10.1177/1071100717735074. Epub 2017 Oct 16. PMID 29035584
- [Background] 8-Eichenholtz SN. Charcot Joints. Springfield, IL, USA: Charles C. Thomas; 1966.
- [Background] Brodsky JW. Management of Charcot joints of the foot and ankle in diabetes. Semin Arthroplasty. 1992; 3: 58-62.
- [Background] Brodsky JW. Patterns of breakdown in the Charcot tarsus of diabetics and relation to treatment. Foot and Ankle 1986;5:353.
- [Background] Lowery NJ, Woods JB, Armstrong DG, Wukich DK. Surgical management of Charcot neuroarthropathy of the foot and ankle: a systematic review. Foot Ankle Int. 2012 Feb;33(2):113-21. doi: 10.3113/FAI.2012.0113. PMID 22381342
- [Background] Anthony S., Pomeroy G. (2016) Exostectomy for Charcot Arthropathy. In: Herscovici, Jr. D. (eds) The Surgical Management of the Diabetic Foot and Ankle. Springer, Cham
- [Background] Tan E.W., Schon L.C. (2016) Plate Fixation Techniques for Midfoot and Forefoot Charcot Arthropathy. In: Herscovici, Jr. D. (eds) The Surgical Management of the Diabetic Foot and Ankle. Springer, Cham
- [Background] Use of External Fixation for the Management of the Diabetic Foot and AnkleDO - 10.1007/978-3-319-27623-6_13 - The Surgical Management of the Diabetic Foot and Ankle
- [Background] Clinics in podiatric medicine and surgery, ISSN: 1558-2302, Vol: 34, Issue: 2, Page: 275-280 .2017
- [Background] Gentili A, Masih S, Yao L, Seeger LL. Pictorial review: foot axes and angles. Br J Radiol. 1996 Oct;69(826):968-74. doi: 10.1259/0007-1285-69-826-968. PMID 9038535
- [Background] Kitaoka HB, Alexander IJ, Adelaar RS, Nunley JA, Myerson MS, Sanders M. Clinical rating systems for the ankle-hindfoot, midfoot, hallux, and lesser toes. Foot Ankle Int. 1994 Jul;15(7):349-53. doi: 10.1177/107110079401500701. PMID 7951968
- [Background] 18-Abetz L, Sutton M, Brady L, McNulty P, Gagnon DD. The diabetic foot ulcer scale (DFS): a quality of life instrument for use in clinical trials. Prac Diabetes Int. 2002;19:167-175.
- [Result] Robinson AH, Pasapula C, Brodsky JW. Surgical aspects of the diabetic foot. J Bone Joint Surg Br. 2009 Jan;91(1):1-7. doi: 10.1302/0301-620X.91B1.21196. PMID 19091997